Physical therapy treatment once a month versus once a week for posture improvement in children and adolescents

Document Date: October 31, 2016

**Clinical Trials NCT03046472** 

## Statistical Plan

Dependent Variables: Thorax Curve Angle, Postural behavior, LBP

Independent Variables: Demographic variables, study groups

## Statistical analysis plan

To compare categorical and dichotomist independent variables we will use  $^2\chi$  - test.

To compare consecutive independent variables we will use t – test.

To compare between frequencies of treatment (two groups) on Thorax Curve Angle and LBP we will use 2 - way ANOVA test.

To compare between frequencies of treatment (two groups) on postural behavior we will use 2 - way ANOVA test. If variables will not distribute normally, we will use a-parametric test.

A Multiple Linear Regression will be used to measure the influence on consecutive dependent variables (VAS for example), and a Logistic Regression for multiple variables will be used to measure the influence on categorical and dichotomist ones.